CLINICAL TRIAL: NCT06817655
Title: Implementation and Evaluation of Peer Support in Oncology in France : a Multisite Participatory Action Research - Adaptation and Transfer in France of the Quebec PAROLE ONCO Research Program
Brief Title: The Research of French PaRole OncO : A Peer Supported Program for Cancer Patients
Acronym: PROOF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL23_1301
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Peer support; Cancer; participatory research; Patient advisor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention consists of patient accompaniment by patient advisors. At least one patient advisor is recruited in each service participating in the study. Patients will be paired with patient advisor and can benefit from accompaniment during their hospital stays or remotely (by phone). The patient advisor will, in turn, be supported by the healthcare professionals' team as well as through a community of practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (PaRole OncO France program) (Experimental): Patients participate in the PaRole OncO France program for which they are matched with a patient advisor and followed throughout treatment in person and/or phone.
  Interventions: Behavioral: PaRole OncO France : Individual peer support

INTERVENTIONS:
Behavioral: PaRole OncO France : Individual peer support — Following the development of the peer support program "PaRole OncO France", we are now proceeding with its implementation and evaluation through a pilot study. This study aims to derive both implementation-related and clinically relevant results.
  Prior to their assignment, all peer helpers undergo a comprehensive training course to ensure they are well-equipped for their role.
  Patients receive individual peer support during their treatment visits, providing real-time assistance and support within the clinical setting.
  The study incorporates three key measurement time points:
  1. Baseline measurement (before the intervention)
  2. After the intervention
  3. Follow-up measurement (1months after the first intervention)
  4. Follow-up measurement (6 months after the first intervention)
  At each time points, participants will complete a set of standardized questionnaires. These instruments are designed to capture relevant outcomes and experiences related to the peer support intervention.

SUMMARY:
Peer support is a valuable mode of accompaniment between individuals who are facing or have faced similar challenging life experiences. In this context, a patient advisor (PA) shares their experiential knowledge, derived from living with a disease, to offer emotional, experiential, and informational support to other patients. This PA intervention represents an innovative form of support for oncology patients, potentially addressing their needs more comprehensively throughout the care pathway by integrating psychosocial dimensions into the support approach.

The present pilot study aims to investigate the implementation and effectiveness of the peer-to-peer support program "PaRole OncO France" in the oncology setting. The study will focus on:

1. Evaluating clinical and psychosocial parameters
2. Utilizing an in-depth multiple case study approach This research seeks to provide insights into how peer support can enhance the overall care experience for oncology patients, potentially leading to improved patient outcomes and a more holistic approach to cancer care.

DETAILED DESCRIPTION:
Peer support is a valuable mode of accompaniment between individuals who are facing or have faced similar challenging life experiences. In this context, a patient advisor (PA) shares their experiential knowledge, derived from living with a disease, to offer emotional, experiential, and informational support to other patients. This PA intervention represents an innovative form of support for oncology patients, potentially addressing their needs more comprehensively throughout the care pathway by integrating psychosocial dimensions into the support approach.

The present pilot study aims to investigate the implementation and effectiveness of the peer-to-peer support program "PaRole OncO France" in the oncology setting. The study will focus on:

1. Evaluating clinical and psychosocial parameters
2. Utilizing an in-depth multiple case study approach This research seeks to provide insights into how peer support can enhance the overall care experience for oncology patients, potentially leading to improved patient outcomes and a more holistic approach to cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants :

  * Patients with newly diagnosed or recurrent cancer (urological, digestive, mammary, pulmonary, ORL, peritoneal carcinosis, melanoma, oncohaematology)
  * French-speaking patients
* Patients adivsors :

  * Patient advisors will be past cancer patients not currently undergoing treatment for their cancer, and considered without evidence of disease
  * French-speaking patients

Exclusion Criteria:

* Patients participants :

  * Not followed in one of the participating units
  * Persons deprived of their liberty by judicial or administrative decision
  * Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Patient advisors :

  * Recurrence of the disease
  * Currently undergoing treatment for active cancer

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementation of the Peer Support Program in Oncology | 30 months
  Acceptability of PH intervention by patients, professionals, and PAs Number of PHs integrated per unit Maintenance of PH activity during the study period in each unit Primary outcome measure is multidimensional by design, as the evaluation of a peer support program requires simultaneous analysis of complementary aspects (acceptability, feasibility, fidelity). These elements are inherently interconnected within our methodological framework.

SECONDARY OUTCOMES:
Evolution of stress levels | Baseline
  Hospital Anxiety and Depression Scale (Min: 0; Max: 42). Higher scores indicate levels of anxiety and depression
Evolution of stress levels | 6 months
  Hospital Anxiety and Depression Scale ((Min : 0; Max : 42).Higher scores indicate greater levels of anxiety and depression.
Evolution of quality of life | Baseline
  EORTC QLQ-C30 questionnaire(Min : 0 ; Max : 100).Higher scores indicate better health status and quality of life
Evolution of quality of life | 1 month, 6 month
  EORTC QLQ-C30 questionnaire(Min : 0 ; Max : 100).Higher scores indicate better health status and quality of life.
Evolution of patient-perceived care experience | Baseline
  Picker Patient Experience questionnaire(Min : 0 ; Max : 100).Higher scores indicate a better patient experience and greater satisfaction.
Evolution of patient-perceived care experience | 1 month
  Picker Patient Experience questionnaire(Min : 0 ; Max : 100).Higher scores indicate a better patient experience and greater satisfaction.
Evolution of patient-perceived care experience | 6 months
  Picker Patient Experience questionnaire(Min : 0 ; Max : 100). Higher scores indicate a better patient experience and greater satisfaction.
Patient empowerment | Baseline
  CASE-cancer questionnaire(Min :0 ; Max : 100). Higher scores indicate greater self-efficacy in managing cancer.
Patient empowerment | 1 month
  CASE-cancer questionnaire(Min :0 ; Max : 100). Higher scores indicate greater self-efficacy in managing cancer.
Patient empowerment | 6 month
  CASE-cancer questionnaire(Min :0 ; Max : 100). Higher scores indicate greater self-efficacy in managing cancer.
Evolution of relationship between accompanied patients and healthcare professionals | Baseline;1 month and 6 month after intervention
  CADICEE questionnaire(Min :0 ; Max : 100). Higher scores indicate a better perception of patient-healthcare partnership
Evolution of quality of life of patient advisors | Baseline, 1month, 6 month
  SF-12 questionnaire(Min :0 ; Max : 100)Higher scores indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No